CLINICAL TRIAL: NCT01774123
Title: Optical Coherence Tomography in Multiple Sclerosis Patients
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Peter Kaiser, Principal Investigator, The Cleveland Clinic
Other Study IDs: 12-422
Record Dates: First submitted 2012-09-17; First posted 2013-01-23 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Multiple Sclerosis; Optic Neuritis
MeSH Terms: conditions — Multiple Sclerosis; Optic Neuritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy: Healthy controls
- MS-ON: Multiple sclerosis with optic neuritis
- MS-NON: Multiple sclerosis without optic neuritis

SUMMARY:
To evaluate the ability of different spectral domain optical coherence tomography (OCT) devices, as well as different acquisition and analysis packages, to detect disease progression in patients with multiple sclerosis with and without a history of optic neuritis

DETAILED DESCRIPTION:
Optical coherence tomography imaging of the retina has been shown to be an effective non invasive method to study retinal changes associated with multiple sclerosis induced optic neuritis. The retina is a unique structure in that it is an unmyelinated part of the central nervous system (CNS). However, it is uncertain which layer of the retina provides the best correlation with MS disease. The investigators propose a prospective, case-control study to compare OCT measurements from different parts of the retina of MS patients with optic neuritis, those without optic neuritis, and healthy controls. The investigators will then correlate the OCT measurements to clinical measures of disease. This will allow future studies to use OCT technology as a primary outcome in studying MS axonal and cell body injury of the CNS, as well as evaluating strategies in treating MS.

ELIGIBILITY:
Inclusion criteria (MS with acute optic neuritis group):

* History of unilateral optic neuritis as a manifestation of multiple sclerosis.
* Age between 18 and 65, inclusive.
* Ability to perform adequate OCT exam.
* Able to provide informed consent to participate in study.

Exclusion criteria (MS with acute optic neuritis group):

- Refractive error greater than ±6 diopters.

Inclusion criteria (MS without acute optic neuritis group):

* History of multiple sclerosis without optic neuritis
* Age between 18 and 65, inclusive.
* Ability to perform adequate OCT exam.
* Able to provide informed consent to participate in study.

Exclusion criteria (MS without acute optic neuritis group):

- Refractive error greater than ±6 diopters.

Inclusion criteria (healthy controls):

* Age between 18 and 65, inclusive.
* Ability to perform adequate OCT exam.
* Able to provide informed consent to participate in the study.

Exclusion criteria (healthy controls):

* Prior history of neurological disease.
* First degree relative with MS.
* Refractive error greater than ±6 diopters.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prospective, case-control study of patients from the Mellen Center and Cole Eye Institute of the Cleveland Clinic in Cleveland Ohio. The study population will consist of MS patients with a prior history optic neuritis in one eye. The affected eye will serve as cases for the study. The contralateral, unaffected eye will be used as the control. Controls will also be recruited from MS patients without a history of optic neuritis and from healthy individuals from Cole Eye Institute.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Thickness of retinal layer | 1 day
  The primary outcome is to determine the thickness of the retinal layers (measured in microns) of optic neuritis-affected eye in MS patients, as compared to controls.

SECONDARY OUTCOMES:
Iris area | 1 day
  Determine the area of the iris (measured in square microns) of optic neuritis-affected eye in MS patients, as compared to controls.

CONTACTS AND LOCATIONS:
Overall Officials: Peter K. Kaiser, MD, Principal Investigator — Cleveland Clinic Cole Eye Institute; Robert Bermel, MD, Principal Investigator — Cleveland Clinic Mellen Center
Locations (1):
- Cole Eye Institute, Cleveland, Ohio, United States

REFERENCES:
- [Background] Frohman EM, Fujimoto JG, Frohman TC, Calabresi PA, Cutter G, Balcer LJ. Optical coherence tomography: a window into the mechanisms of multiple sclerosis. Nat Clin Pract Neurol. 2008 Dec;4(12):664-75. doi: 10.1038/ncpneuro0950. PMID 19043423
- [Background] Siger M, Dziegielewski K, Jasek L, Bieniek M, Nicpan A, Nawrocki J, Selmaj K. Optical coherence tomography in multiple sclerosis: thickness of the retinal nerve fiber layer as a potential measure of axonal loss and brain atrophy. J Neurol. 2008 Oct;255(10):1555-60. doi: 10.1007/s00415-008-0985-5. Epub 2008 Sep 25. PMID 18825432